CLINICAL TRIAL: NCT01115530
Title: An Exercise and Nutritional Intervention for Deconditioned Older Adults
Brief Title: Exercise and Nutritional Intervention for Deconditioned Older Adults
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient subject recruitment.
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7142-R
Record Dates: First submitted 2010-02-25; First posted 2010-05-04 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Muscle Weakness
MeSH Terms: conditions — Muscle Weakness | interventions — Resistance Training; Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (No Intervention): Control inpatient GEM rehabilitation and continue twice weekly low level walking/stretching to control for time/interaction with intervention/exercise groups
- 2 (Experimental): Resistance exercise (2x/week)
  Interventions: Other: Resistance exercise
- 3 (Experimental): Nutritional (amino acid metabolite) supplement twice daily
  Interventions: Dietary Supplement: Protein and HMB (see below) supplement
- 4 (Experimental): Resistance exercise (2x/week) and nutritional (amino acid metabolite) supplement twice daily
  Interventions: Other: Resistance exercise; Dietary Supplement: Protein and HMB (see below) supplement

INTERVENTIONS:
Other: Resistance exercise — Lower extremity resistance exercise (leg press/knee extension) twice per week for 12 weeks
  Arms: 2; 4
Dietary Supplement: Protein and HMB (see below) supplement — Ingested twice daily for 12 weeks Active components include: Protein and B-hydroxy-B -methylbutyrate
  Arms: 3; 4

SUMMARY:
In this study we will evaluate whether the addition of a formal lower extremity resistance exercise training program and/or a nutritional supplement will improve the functional recovery of older adult veterans participating in a geriatric rehabilitation program for deconditioning. Specifically, subjects admitted to a geriatric inpatient rehabilitation program with a diagnosis of deconditioning will be randomly assigned to one of four groups; 1) Control/standard rehabilitation program, 2) Standard rehabilitation plus resistance exercise twice per week, 3) Standard rehabilitation plus a daily nutritional supplement, 4) Standard rehabilitation plus the resistance exercise and the nutritional supplement. Subjects will participate in each program for 12 weeks. At the beginning and end of the study we will measure lower extremity strength, walking speed, and overall function (using the standardized Functional Independence Measure), and compare the changes in each group.

ELIGIBILITY:
Inclusion Criteria:

* Veteran admitted to GEM rehabilitation unit
* Primary problem: Deconditioning/Generalized Weakness
* Age 65-90
* Self reported ability to report to the CAVHS GRECC twice per week after discharge from the GEM unit.
* Living in the community prior to recent acute care hospitalization
* Decision making capacity to be able to consent to the study as documented in the GEM attending or GEM APN's admission note

Exclusion Criteria:

* Conditions that are exclusionary criteria for GEM admission including the following: direct transfer from any ICU, end-stage chronic medical/surgical disorder with no rehabilitation potential, terminal diagnosis /hospice/respite care, hemodialysis, active radiation therapy. Also, Type I diabetes mellitus
* Any other condition considered exclusionary by the PI / study physician.

Prior to group assignment, subjects will be evaluated for contraindications to exercise training per the American College of Sports Medicine (ACSM)guidelines including the following:

* Myocardial infarction documented in the past 3 months
* Unstable angina (at rest in past 3 months, or increased angina pattern in past month)
* Uncorrected left main coronary obstruction > 50%;
* Congestive heart failure exacerbation in past 3 months (symptoms at rest or worsening symptoms requiring change in baseline diuretic dose)
* Severe valvular heart disease (aortic or mitral stenosis with valve area < 1 cm2 , mitral or aortic insufficiency with any degree of LV dysfunction, pulmonary hypertension [PASP > 50 mmHg], or LV enlargement [LVESD 40 mm, or LVEDD > 55 mm])
* Active pericarditis / myocarditis
* Malignant or unstable arrhythmias, third degree AV block without pacemaker
* Elevated resting blood pressure (systolic > 200 mmHg, diastolic > 110 mmHg)
* Known large (> 4 cm) aortic aneurysm
* Known cerebral aneurysm or intracranial bleed in past 1 year
* Terminal cancer
* Acute retinal hemorrhage or ophthalmologic surgery within 3 months

Ages: 65 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2012-07 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Function by the Functional Independence Measure | 12 weeks

SECONDARY OUTCOMES:
Gait speed | 12 weeks
Lower extremity strength | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Kortebein, MD, Principal Investigator — Central Arkansas VHS Eugene J. Towbin Healthcare Ctr, Little Rock
Locations (1):
- Central Arkansas VHS Eugene J. Towbin Healthcare Ctr, Little Rock, No. Little Rock, Arkansas, United States